CLINICAL TRIAL: NCT07184658
Title: A Prospective Randomized Controlled Trial of Ultrasound-Guided Repeated Normal Saline Injections for Preventing and Treating Tendon Adhesion
Brief Title: Ultrasound-Guided Multiple Saline Injections for Prevention of Tendon Adhesion: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kai Wang (Other)
Responsible Party: Sponsor-Investigator, Kai Wang, Principal Investigator, Department of Orthopaedics, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-119; 82425035 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-09-18; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Tendon Adhesion
Keywords: Ultrasound-guided injection; Normal saline; Tendon adhesion prevention; Flexor tendon repair; Hand surgery; Randomized controlled trial
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized controlled trial with parallel assignment. Patients undergoing flexor tendon repair will be randomly allocated to either the intervention group (ultrasound-guided saline injections) or the control group (no injection).
Masking Description: This is an open-label study; no masking will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Ultrasound-guided Saline Injection (Experimental): Patients will undergo ultrasound-guided peritendinous injections of 1 mL normal saline at the tendon repair site on postoperative days 7, 14, and 21. The goal is to prevent tendon adhesion and improve functional outcomes.
  Interventions: Procedure: Ultrasound-guided peritendinous saline injection
- Control Group - Standard Care (No Intervention): Patients will receive standard postoperative care after tendon repair without saline injection.

INTERVENTIONS:
Procedure: Ultrasound-guided peritendinous saline injection — Under ultrasound guidance, 1 mL of sterile normal saline will be injected peritendinously at the tendon repair site at 7, 14, and 21 days after surgery to reduce adhesion formation and preserve tendon healing.
  Other Names: Normal saline injection
  Arms: Intervention Group - Ultrasound-guided Saline Injection

SUMMARY:
This prospective randomized controlled trial aims to evaluate the efficacy and safety of ultrasound-guided repeated normal saline injections for the prevention and treatment of tendon adhesion following flexor tendon repair. Tendon adhesion is a common complication after tendon injury, leading to pain, stiffness, and impaired hand function. Conventional anti-adhesion strategies, such as physical barrier membranes, may induce local inflammation or have limited effectiveness.

In this study, patients undergoing tendon repair will be randomly assigned to receive either ultrasound-guided peritendinous saline injections at 7, 14, and 21 days after surgery (intervention group) or no injection (control group). The primary outcome is total active motion (TAM-%) at 3 months after surgery. Secondary outcomes include TAM-% at 6 weeks, pain scores (VAS), Michigan Hand Questionnaire (MHQ) scores, infection rate, and tendon rupture rate. A total of 136 patients will be enrolled (68 in each group).

The findings of this trial will help to establish whether repeated saline injections under ultrasound guidance can effectively prevent tendon adhesion, improve pain and functional outcomes, and ensure tendon healing with minimal complications.

DETAILED DESCRIPTION:
Tendon adhesion is one of the most common complications following flexor tendon repair, with an incidence of up to 60%. Adhesion significantly impairs hand function, often leading to a cycle of adhesion formation, surgical release, and recurrent adhesion, which causes long-term disability and high healthcare costs. Current preventive measures mainly rely on physical barrier materials, such as membranes or gels, but these approaches may induce aseptic inflammation and pain, and their long-term effectiveness remains limited.

Our previous research suggested that early peritendinous injection therapy may be more effective than intraoperative application in preventing tendon adhesion. Using dynamic ultrasound, we successfully localized tendon adhesion sites and demonstrated the feasibility of delivering precise peritendinous injections under ultrasound guidance. Based on these findings, we hypothesize that repeated ultrasound-guided saline injections at early postoperative stages can reduce adhesion formation while minimizing the impact on tendon healing.

This is a prospective, single-center, randomized controlled clinical trial enrolling 136 patients (68 per group) after flexor tendon repair. Patients in the intervention group will undergo ultrasound-guided peritendinous injections of 1 mL normal saline on postoperative days 7, 14, and 21. The control group will receive standard care without injections. Patients will be followed up at 6 weeks and 3 months after surgery. The primary endpoint is total active motion (TAM-%) at 3 months. Secondary endpoints include TAM-% at 6 weeks, visual analog scale (VAS) pain scores, Michigan Hand Questionnaire (MHQ) scores, infection rate, tendon rupture rate, and wound healing time.

Safety will be assessed through physical examinations, laboratory tests (blood count, C-reactive protein, erythrocyte sedimentation rate), and adverse event monitoring. Statistical analysis will be performed using appropriate parametric or non-parametric methods, with significance set at P < 0.05.

The successful completion of this study is expected to provide clinical evidence supporting ultrasound-guided saline injections as a safe, effective, and low-cost strategy for preventing tendon adhesion, improving hand function, and reducing complications.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 60 years. Diagnosed with flexor tendon rupture. Scheduled for surgical tendon repair.

Exclusion Criteria:

Associated vascular or nerve injury. History of diabetes mellitus. History of non-steroidal anti-inflammatory drug (NSAID) treatment. History of cardiac insufficiency. History of hematologic diseases. History of hepatic or renal dysfunction. History of rheumatologic or autoimmune diseases. History of radiotherapy or chemotherapy. History of corticosteroid treatment. Pregnancy. Currently participating in another clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Total Active Motion Percentage (TAM-%) of the injured finger at 3 months after surgery | 3 months after tendon repair
  TAM-% is calculated as the sum of active flexion at the metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints minus the sum of extension deficits, divided by the normal range of motion, multiplied by 100%. It reflects functional recovery and tendon adhesion severity.

SECONDARY OUTCOMES:
Pain score (VAS) | 6 weeks and 3 months after surgery
  Visual Analog Scale (0-10), where 0 = no pain and 10 = worst imaginable pain.
TAM-% at 6 weeks after surgery | 6 weeks after tendon repair
  Same calculation method as the primary outcome, evaluated at an earlier time point.
Michigan Hand Questionnaire (MHQ) score | 3 months after surgery
  Patient-reported outcome measure assessing hand function, activities of daily living, pain, work performance, aesthetics, and satisfaction.
Tendon rupture rate | Within 3 months after surgery
  Incidence of tendon rupture confirmed by clinical examination or imaging.
Infection rate | Within 3 months after surgery
  Incidence of superficial or deep surgical site infections diagnosed according to clinical and laboratory criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Shen LIU, MD, Principal Investigator — Shanghai 6th Peoples Hospital Affiliated to Shanghai Jiaotong University School of Medicine Department of Orthopaedic Surgery
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared due to concerns regarding patient privacy and institutional regulations.

REFERENCES:
- [Background] Franssen AJPM, Degens JHRJ, Daemen JHT, Laven IEWG, Hulsewe KWE, Vissers YLJ, de Loos ER. Mediastinal staging by thoracic surgeons: are we close to a paradigm shift? J Thorac Dis. 2023 Jan 31;15(1):10-13. doi: 10.21037/jtd-22-1420. Epub 2023 Jan 6. No abstract available. PMID 36794129
- [Background] Ockun MA, Gercek YC, Demirsoy H, Demirsoy L, Macit I, Oz GC. Comparative evaluation of phenolic profile and antioxidant activity of new sweet cherry (Prunus avium L.) genotypes in Turkey. Phytochem Anal. 2022 Jun;33(4):564-576. doi: 10.1002/pca.3110. Epub 2022 Feb 4. PMID 35122339
- [Background] Yasmeen R, Zahid B, Alyas S, Akhtar R, Zahra N, Kouser S, Hashmi AS, Athar M, Tayyab M, Anjum AA. Ameliorative effects of Lactobacillus against Aflatoxin B1. Braz J Biol. 2021 Dec 20;84:e250517. doi: 10.1590/1519-6984.250517. eCollection 2021. PMID 34932626
- [Background] Sueiras M, Sahuquillo J, Garcia-Lopez B, Sanchez-Guerrero A, Poca MA, Santamarina E, Riveiro M, Fabricius M, Strong AJ. [Cortical spreading depolarization phenomena in patients with traumatic and ischemic brain injuries. Results of a pilot study]. Med Intensiva. 2014 Oct;38(7):413-21. doi: 10.1016/j.medin.2013.09.008. Epub 2013 Dec 15. Spanish. PMID 24342071
- [Background] Roy V, Sahni P, Gupta P, Sethi GR, Khanna A. Blood levels of pyrazinamide in children at doses administered under the Revised National Tuberculosis Control Program. Indian Pediatr. 2012 Sep;49(9):721-5. doi: 10.1007/s13312-012-0164-8. Epub 2011 Jan 17. PMID 22317983
- [Background] Kim HT, Oh JS, Lee JS, Lee TH. Z-lengthening of the Achilles tendon with transverse skin incision. Clin Orthop Surg. 2014 Jun;6(2):208-15. doi: 10.4055/cios.2014.6.2.208. Epub 2014 May 16. PMID 24900904
- See also: Related Info — https://www.shsmu.edu.cn/english/info/1085/1228.htm